CLINICAL TRIAL: NCT01036841
Title: Influence of Food-intake on Pharmacokinetic and Pharmacodynamic Parameters of Desmopressin Oral Tablet Formulation, in Comparison With Desmopressin MELT Formulation
Brief Title: Influence of Food-intake on Desmopressin Oral Tablets and MELT-formulation
Acronym: TM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009/653
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Enuresis; Polyuria
Keywords: MNE with nocturnal polyuria; monosymptomatic nocturnal enuresis with nocturnal polyuria
MeSH Terms: conditions — Enuresis; Polyuria | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- desmopressin tablet (Active Comparator)
  Interventions: Drug: desmopressin tablet
- desmopressin MELT-formulation (Experimental)
  Interventions: Drug: desmopressin MELT formulation

INTERVENTIONS:
Drug: desmopressin tablet — Administration of desmopressine tablet
  Arms: desmopressin tablet
Drug: desmopressin MELT formulation — Administration of desmopressine MELT formulation
  Arms: desmopressin MELT-formulation

SUMMARY:
Alarm-treatment as well as Desmopressin, a synthetic analogue of human vasopressin, are considered the only evidence-based medicine (EBM) IA treatments in monosymptomatic nocturnal enuresis (MNE). Desmopressin exists in three different formulations for ambulant use: nasal spray, tablet and lyophilisate (MELT) each with differences in bioavailability (spray 2%, tablet 0.2%, MELT 0.5%). There 's insufficient evidence to confirm the actually used bioequivalent doses ( 10µg spray = 120µg MELT= 0.2mg tablet).

Although so frequently used, very few pharmacokinetic and -dynamic data on desmopressin are available for children.

Due to prolonged half life, associated with waterintoxication,the nasal spray has a black box warning from the FDA and is no longer recommended . For some authors oral formulations appear to be a safer alternative. However, based on clinical experience of less response rate with oral formulations, lower biodisponibility is suspected. Adult research confirms low bioavailability of tablets but also show major influences by food-intake and changes in gastro-intestinal motility.

To achieve maximum efficacy, recommendations are to take desmopressin tablet 1 hour before bedtime and 2 hours after meal: this is unrealistic in schoolaged children since there never is 3 hours between evening meal and bedtime.

In 2005 a dose response study demonstrated superior pharmaco-kinetic and dynamic properties for desmopressin Lyophilisate MELT formula.

Since these results implicate superior action of MELT, often a change to MELT is recommended if there is a suboptimal response with tablet: sublingual absorption would eliminate the influence of food-intake.

However, for this statement there's no evidence, since these tests were all conducted in children in fasting condition. Only one clinical study demonstrates bioequivalence for MELT and tablet.

Hypothesis is that desmopressin MELT formulation has a better bioavailability when administered together with meal due to its sublingual absorption.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-16 years old
* with MNE and nocturnal polyuria
* treated with desmopressin tablet, non or partial responders, for whom change to MELT formulation is indicated according to the international standard guidelines.

Exclusion Criteria:

* history of urologic disease, diurnal urinary incontinence, diabetes insipidus, urinary tract infection, clinically significant disease
* No systemic use of antibiotics, diuretics, other medication that influences urinary concentrating mechanism
* abnormalities of oral mucosa which could influence drugrelease or absorption

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Bioavailability of desmopressine MELT and tablet when taken with meal. | at 1h, 2h and 6h post adminstration

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic for desmopressine MELT and tablet. | at 1h, 2h, 3h, 6h and 8h post administration

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vande Walle, MD, PhD, Principal Investigator — University Hospital Ghent, department of pediatric nephrology
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be